CLINICAL TRIAL: NCT00011011
Title: A Randomized Phase I/II Pilot Study of Intermittent Withdrawal of Antiretroviral Therapy as an Immunization Strategy and Double-Blinded Immunization With ALVAC-HIV vCP1452 in Subjects With Persistent CD4+ Cell Counts Greater Than 400 Cells/mm3 and Plasma HIV-1 RNA Levels Less Than 50 Copies/ml
Brief Title: Vaccine (ALVAC-HIV vCP1452) Use and Intermittent Withdrawal of Anti-HIV Drugs in Patients With HIV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: A5068; 10072 (Registry Identifier: DAIDS ES Registry Number); Substudy AACTG A5101s; Substudy AACTG A5111s; Substudy AACTG A5137s; ACTG A5068; AACTG A5068
Record Dates: First submitted 2001-02-08; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Administration Schedule; AIDS Vaccines; CD4 Lymphocyte Count; RNA, Viral; Anti-HIV Agents; Viral Load; HIV Therapeutic Vaccine; Treatment Interruption
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: ALVAC(2)120(B,MN)GNP (vCP1452)

SUMMARY:
Long-term control of HIV depends on improvement in an individual's immune system. The purpose of this study is to see if either stopping anti-HIV drugs for short periods of time and/or adding a vaccine to the anti-HIV drugs being taken will help to better control HIV infection. The study will test whether these treatment approaches are safe. The HIV vaccine in this study has been tested in people who did not have HIV infection and improved the way their immune system worked. This study will evaluate whether these same immune system changes happen in people with HIV, and, if such changes do occur, assess whether these changes help to improve control of HIV in these patients.

DETAILED DESCRIPTION:
The best hope for long-term control of HIV infection in an individual likely rests with the resumption of effective HIV-specific immune responses. Intermittent antiretroviral therapy (ART) withdrawal, as an attempt to "immunize" the subject with his/her own active viral quasi-species population, represents an alternative approach to traditional immunization strategies. This study hopes to determine whether intermittent ART withdrawal serves to stimulate HIV-specific immune responses and control of viral replication. This approach will be compared with vaccination with ALVAC-HIV vCP1452. In addition, it is conceivable that intermittent ART withdrawal could boost and broaden the prime response to exogenous vaccine; that will also be studied.

Patients will continue receiving their potent ART (not provided by the study) and will be randomly assigned to one of four treatment strategies as follows:

Arm A: ALVAC placebo and potent ART for 92 weeks with a single 12- to 20-week therapy withdrawal period; Arm B: ALVAC placebo and potent ART for 84 weeks with a 4- to 6-week therapy withdrawal period, a 4-week therapy withdrawal period, and a 12- to 20-week therapy withdrawal period; Arm C: ALVAC vCP1452 vaccine and potent ART for 92 weeks with a single 12- to 20-week therapy withdrawal period; and Arm D: ALVAC vCP1452 vaccine and potent ART for 84 weeks with a 4- to 6-week therapy withdrawal period, a 4-week therapy withdrawal period, and a 12- to 20-week therapy withdrawal period.

Immunizations of placebo or vaccine wil be administered in 3 separate sets of 3 injections per set (9 total) and immunization schedules are the same for all patients, those undergoing intermittent therapy withdrawal (Arms B and D) and those who are not (Arms A and C).

This is a multiple-step study. Patients in Arms B and D will receive a 4-week period of potent ART therapy along with the first set of immunizations (Step 1) followed by therapy withdrawal for 4 to 6 weeks (Step 2). Alternating periods of therapy resumption (Step 3, consisting of 16 weeks on potent ART with the second set of vaccine administrations), a second therapy withdrawal (Step 4 for 4 weeks), and another therapy resumption (Step 5, consisting of 16 weeks on potent ART with the third set of vaccine administrations) will follow. Patients in Arms A and C will remain on Step 1 for the first 44 weeks on study.

After 44 to 46 weeks on study, patients in all arms will have therapy withdrawn for 12 to 20 weeks (Step 6). Following completion of Step 6, patients whose viral load are below 10,000 copies/ml will be encouraged to remain off potent ART (Step 7) until completion of the study, as long as CD4 T-cell levels remain 50 percent or more of their baseline levels. Participants who successfully complete Step 7 will be invited to enter Step 9, a 48-week optional protocol extension. Otherwise, patients will restart their potent ART regimens (Step 8) and receive virologic and CD4 T-cell monitoring until completion of the study.

All patients will be monitored at regular clinic visits. Viral load and CD4 T-cell counts will be measured at each visit. Patients in all arms may participate in substudy A5101s (Male Genital Secretions) or substudy A5137s (Female Genital Secretions), and patients in Arms B and D may participate in substudy A5111s (Latent Infected T-Cell Clearance).

ELIGIBILITY:
Inclusion Criteria for Step 1

* HIV infection
* CD4 count greater than 400 cells/mm3 within 6 months before study entry
* Current, persistent viral load below 400 copies/ml for 6 months before study entry and under 50 copies/ml at study screening
* Currently receiving their first combination ART regimen (3 or more antiretrovirals) for at least 4 weeks before screening, or if the current potent ART regimen is not their first potent ART regimen, must have been receiving the current regimen for at least 4 weeks prior to screening
* Negative pregnancy test within 45 days before study entry
* Acceptable methods of contraception
* Provide informed consent

Exclusion Criteria

* Immunomodulators within 45 days of study entry such as systemic corticosteroids, interferons, interleukins, thalidomide, sargramostim (granulocyte-macrophage colony-stimulating factor [GM-CSF]), dinitrochlorobenzene (DNCB), thymosin alpha, thymopentin, inosiplex, polyribonucleoside, and ditiocarb sodium
* Abacavir within 8 weeks of study entry
* Infection or medical illness within 14 days of study entry
* Cancer that may require systemic therapy
* History of lymph node radiation therapy
* Prior HIV vaccine
* Received hydroxyurea within 45 days of study entry
* Close contact with canaries through work (e.g., breeding farms, bird shops); patients with a pet canary are not excluded
* Abuse or dependence on drugs or alcohol
* Allergic to albumin
* Pregnant or breastfeeding
* Infected with HIV within 1 year of study entry
* Interruption of potent ART for more than 7 consecutive days within 1 year of study entry
* History of allergy to egg proteins or neomycin
* History of other serious acute allergic reactions (e.g., anaphylaxis, allergy-induced asthma, Stevens-Johnson syndrome, toxic epidermal necrolysis)

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2001-02; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M. Jacobson, MD, Study Chair — Beth Israel Medical Center; Ian Frank, MD, Study Chair — Division of Infectious Diseases, University of Pennsylvania
Locations (16):
- United States (16):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - UCLA CARE Center CRS, Los Angeles, California
  - Ucsf Aids Crs, San Francisco, California
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Washington U CRS, St Louis, Missouri
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - AIDS Care CRS, Rochester, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Case CRS, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - Univ. of Pennsylvania Health System, Presbyterian Med. Ctr., Philadelphia, Pennsylvania
  - The Miriam Hosp. ACTG CRS, Providence, Rhode Island
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Ferrari G, Berend C, Ottinger J, Dodge R, Bartlett J, Toso J, Moody D, Tartaglia J, Cox WI, Paoletti E, Weinhold KJ. Replication-defective canarypox (ALVAC) vectors effectively activate anti-human immunodeficiency virus-1 cytotoxic T lymphocytes present in infected patients: implications for antigen-specific immunotherapy. Blood. 1997 Sep 15;90(6):2406-16. PMID 9310492
- [Background] Rosenberg ES, Billingsley JM, Caliendo AM, Boswell SL, Sax PE, Kalams SA, Walker BD. Vigorous HIV-1-specific CD4+ T cell responses associated with control of viremia. Science. 1997 Nov 21;278(5342):1447-50. doi: 10.1126/science.278.5342.1447. PMID 9367954
- [Background] Belshe RB, Gorse GJ, Mulligan MJ, Evans TG, Keefer MC, Excler JL, Duliege AM, Tartaglia J, Cox WI, McNamara J, Hwang KL, Bradney A, Montefiori D, Weinhold KJ. Induction of immune responses to HIV-1 by canarypox virus (ALVAC) HIV-1 and gp120 SF-2 recombinant vaccines in uninfected volunteers. NIAID AIDS Vaccine Evaluation Group. AIDS. 1998 Dec 24;12(18):2407-15. doi: 10.1097/00002030-199818000-00009. PMID 9875578
- [Result] Jacobson JM, Pat Bucy R, Spritzler J, Saag MS, Eron JJ Jr, Coombs RW, Wang R, Fox L, Johnson VA, Cu-Uvin S, Cohn SE, Mildvan D, O'Neill D, Janik J, Purdue L, O'Connor DK, Vita CD, Frank I; National Institute of Allergy and Infectious Diseases-AIDS Clinical Trials Group 5068 Protocol Team. Evidence that intermittent structured treatment interruption, but not immunization with ALVAC-HIV vCP1452, promotes host control of HIV replication: the results of AIDS Clinical Trials Group 5068. J Infect Dis. 2006 Sep 1;194(5):623-32. doi: 10.1086/506364. Epub 2006 Aug 1. PMID 16897661